CLINICAL TRIAL: NCT02988609
Title: Concussion in Rugby Players: a Pilot Study of Neural Recovery Using Functional Magnetic Resonance Imaging (fMRI)
Brief Title: Concussion in Rugby Players: a Pilot Study of Neural Recovery Using fMRI
Acronym: RugbyCom
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in enrollment and changes in methodology
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/15/7730
Record Dates: First submitted 2016-05-13; First posted 2016-12-09 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concussion Group (Experimental): Players with a recent (<72 hours) history of concussion will be assessed 3 times. just after concussion, after disappearance of clinical symptoms and 3 months after the previous visit. During each visit, participant will undergo a neurological and a neuropsychological assessment and a structural and resting state fMRI.
  Interventions: Device: fMRI
- Control Group (Active Comparator): a control group with no history of concussion will be the comparator. Participants will be assessed 3 times. Visits will be the same for the control group and duration between visits in this group will be matched to the concussion group. During each visit, participant will undergo a neurological and a neuropsychological assessment and a structural and resting state fMRI.
  Interventions: Device: fMRI

INTERVENTIONS:
Device: fMRI — fMRI at 3 different times after concussion: just after concussion (V1), once players have clinically recovered (V2) and 3 months after V2 (V3).

SUMMARY:
This study assess the putative persistence of neural damage using resting state fMRI after concussion in rugby player once they have clinically recovered. The hypothesis is that despite a clinical recovery (absence of symptoms; neurological and neuropsychological examination returned to normal) connectivity map obtained using resting state fMRI are significantly different from a group of control subjects.

DETAILED DESCRIPTION:
Resting state fMRI has shown to be a sensitive tool to assess neural damage after concussion. It seems more sensible than structural MRI including DTI. the study goal will be to assess rugby players using fMRI at 3 different times after concussion: just after concussion (V1), once players have clinically recovered (V2) and 3 months after V2 (V3). The study would specifically like to challenge clinical examination supposed to be normal at V2 to connectivity maps using resting state fMRI preformed at the same time. fMRI performed at V1 and V3 will serve as comparators (respectively very altered at V1 and back to normal at V3).

ELIGIBILITY:
Inclusion Criteria:

* no neurological or psychiatric disease
* recent history of concussion (<3 months) according to the Rugby French Federation criteria.

Exclusion Criteria:

* Inability to be assessed by MRI

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Difference of connectivity maps between the players with concussion and the group control | up to 1 month
  connectivity maps obtained during a 10 minutes resting state fMRI at V2

SECONDARY OUTCOMES:
Difference of connectivity maps between the players with concussion and the group control | up to 3 months
  Connectivity maps obtained during a 10 minutes resting state fMRI at V1 and V3
neuropsychological questionnaire | up to 3 months
  Scores obtained the neuropsychological assessment. Memory, attention and executive functions will be assessed using validated tools.
neurophysiological data | up to 3 months
  Structural imaging data (DTI)

CONTACTS AND LOCATIONS:
Overall Officials: David BRAUGE, MD, Principal Investigator — U H Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smits M, Houston GC, Dippel DW, Wielopolski PA, Vernooij MW, Koudstaal PJ, Hunink MG, van der Lugt A. Microstructural brain injury in post-concussion syndrome after minor head injury. Neuroradiology. 2011 Aug;53(8):553-63. doi: 10.1007/s00234-010-0774-6. Epub 2010 Oct 6. PMID 20924757